CLINICAL TRIAL: NCT02797600
Title: Community Awareness, Resources and Education (CARE II) Project: Project 1
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-10095
Record Dates: First submitted 2015-06-08; First posted 2016-06-13 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer
Keywords: Appalachia
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surveys and Questionnaires; Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, saliva samples, buccal scrapes, oral rinse, tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ARM I: Woman residing in Appalachian counties who have prevalent invasive cervical cancer. Invasive cervical cancer cases participants will include women previously and currently treated for ICC during the past 10 years. Questionnaires will be used to obtain self-reported demographic, behavioral, social, family and medical history, and quality of life data. Biological samples will be collected during a scheduled visit with the research staff.
  Interventions: Behavioral: Questionnaires; Other: Biological Samples
- ARM II: Woman residing in Appalachian counties who are newly diagnosed with invasive cervical cancer(ICC). Newly diagnosed with ICC, and currently being treated for ICC. Questionnaires will be used to obtain Questionnaires will be used to obtain self-reported demographic, behavioral, social, family and medical history, and quality of life data. All biological samples will be collected during a scheduled clinic visit.
  Interventions: Behavioral: Questionnaires; Other: Biological Samples
- ARM III: Healthy controls (women without a diagnosis of any type of cancer. Healthy controls will be women who are coming into one of the participating clinic or physician practice for a routine Pap test. Questionnaires will be used to obtain Questionnaires will be used to obtain self-reported demographic, behavioral, social, family and medical history, and quality of life data. All biological samples will be collected at the time of the clinical Pap smear.
  Interventions: Behavioral: Questionnaires; Other: Biological Samples

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires will be used to obtain self-reported demographic, behavioral, social, family and medical history, and quality of life data. The questions are standardized and taken from either nationally recognized surveys, CARE I surveys, or represent validated survey items.
Other: Biological Samples — All biological samples will be collected at the time of the clinical Pap smear for the controls, and will be collected for the Arm 2 (newly diagnosed) during a scheduled clinic visit. For those individuals in Arm 1, biological samples will be collected during a scheduled visit with the research staff.
  Other Names: specimen collection

SUMMARY:
The study hypothesis is that the increased incidence of cervical cancer observed in Appalachian women over their non-Appalachian counterparts is due in part to inherited and somatic alterations of key components of the Transforming Growth Factor β (TGFβ) signaling pathway.

DETAILED DESCRIPTION:
This project is a case control study that is designed to determine prevalence of inherited polymorphic and somatically acquired variants of key TGF-ß pathway components in a large cohort of Appalachian invasive cervical cancer (ICC) patients compared to healthy Appalachian women. It will be determined whether these genetic alterations contribute individually or in combination with other known environmental (Human Papillomavirus, Epstein-Barr Virus), behavioral (smoking), and social (stress, social networks) risk factors, to the increased susceptibility of Appalachian women to ICC development. Women will be recruited from several clinics and physician practices in West Virginia, Charleston and Appalachia Ohio and Kentucky. Participants will be women residing in these area who are 18 years and older, not pregnant, speak English, not cognitively impaired and able to provide informed consent. There will be three distinct types of women recruited into the study; 1. ARM 1 - previously treated for invasive cervical cancer; 2. ARM 2 - newly diagnosed with invasive cervical cancer; and 3. healthy controls - without a diagnosis of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients previously or newly diagnosed with invasive cervical cancer
* healthy women without a diagnosis of any type of cancer
* English speaking
* Able to provide informed consent, biological and questionnaire data.

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be women residing in Appalachian counties (West Virginia and Appalachia Ohio and Kentucky). There will be three distinct types of women recruited into the study; 1) prevalent invasive cervical cancer cases; 2) newly diagnosed invasive cervical cancer cases; and 3) healthy controls (women without a diagnosis of any type of cancer). Women will be recruited from several clinics and physician practices in Appalachian counties.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Genetic variations in TGFβ ligand and receptor genes and other cancer-associated genes. | Day 1
  The number of participants with genetic variations in TGFβ ligand and receptor genes and other cancer-associated genes with known single nucleotide polymorphisms as determined by direct sequencing and SNP PCR analyses

SECONDARY OUTCOMES:
Environmental, behavioral and socioeconomic risk factors. | Day 1
  The number of participants with various environmental, behavioral and socioeconomic risk factors as assessed by survey data.

CONTACTS AND LOCATIONS:
Overall Officials: Electra Paskett, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu